CLINICAL TRIAL: NCT00938613
Title: A Randomized, Double-Blind, Placebo-Controlled, 3-Way Cross-Over Study to Compare the Relative Efficacy of Budesonide Administered Via CE Budesonide Nasal Solution & Rhinocort Aqua in the Treatment of the Symptoms of AR in an EEC Model
Brief Title: Compare CE-Budesonide Nasal Solution & Rhinocort Aqua in an EEC Study of AR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ligand Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CDX947CT001; P2DS06001
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: SAR
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Budesonide; SBE4-beta-cyclodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Captisol-Enabled Budesonide (Experimental): 32 ug/spray
  Interventions: Drug: Budesonide
- Rhinocort Aqua (Active Comparator): 32 ug/spray
  Interventions: Drug: Budesonide
- Placebo (Placebo Comparator): posphate buffered saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide — nasal spray, one spray per nostril at time 0
  Other Names: CDX947; Captisol
  Arms: Captisol-Enabled Budesonide
Drug: Placebo — nasal spray, one spray per nostril at time 0
  Other Names: phosphate buffered saline solution
  Arms: Placebo
Drug: Budesonide — nasal spray, one spray per nostril at time 0
  Other Names: Rhinocort Aqua
  Arms: Rhinocort Aqua

SUMMARY:
The primary objective of this study was to compare the relative efficacy of Budesonide administered via Captisol-Enabled Budesonide nasal solution and Rhinocort Aqua in patients with seasonal allergic rhinitis (SAR) exposed to controlled ragweed pollen using an EEC model.

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Single-Center, Three-Way Cross-Over Study to Compare the Relative Efficacy of Budesonide administered via Captisol-Enabled® Budesonide Nasal Solution and Rhinocort Aqua® (32 µg/spray) in the Treatment of the Symptoms of Allergic Rhinitis in an Environmental Exposure Chamber (EEC).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a clinical history of SAR
* Adults (males and females) aged 18 to 65, inclusive
* Patients must have documentation of a positive skin test within 12 months of screening to ragweed allergen
* Non-pregnant, non-lactating females, or women who are post-menopausal or are naturally or surgically sterile. Females of childbearing potential must have a confirmed absence of pregnancy and must be using an acceptable birth control method
* In generally good health
* Willingness to attend all study visits
* Capable of following and understanding instructions
* Willing and able to provide written informed consent prior to initiation of any study procedures, including initiation of washout of any concomitant medications

Exclusion Criteria:

* Pregnancy, nursing, or plans to become pregnant or donate gametes
* Have clinically significant physical findings of nasal anatomical deformities causing greater than 50% obstruction
* Previous participation in a budesonide study within three months prior to the Screening Visit.
* Participation in any investigational drug trial within the 30 days preceding the Screening Visit, and thereafter.
* A known hypersensitivity to any corticosteroid or any of the excipients in the formulation of the investigational drug
* History of severe respiratory infection or disorder
* History of alcohol or drug abuse
* History of a positive test for HIV, hepatitis B or hepatitis C.
* Active asthma requiring treatment with inhaled or systemic corticosteroid and/or routine use of ß-agonists or any controller drugs, intermittent use (less than or equal to 3 uses per week) of inhaled short acting ß-agonists is acceptable.
* Use of any of the prohibited medications within the identified exclusion periods
* Use of antibiotic therapy for acute conditions within 14 days prior to the Screening Visit and thereafter. Low doses of antibiotics taken for prophylaxis are permitted based on the judgment of the Investigator if therapy was started prior to the Screening Visit AND is expected to continue throughout the study.
* Initiation of immunotherapy or dose escalation during the study period. However, patients may be considered for inclusion if the immunotherapy was initiated 90 days or more prior to the Screening Visit AND if the dosing was stable (maintenance dose) for 30 days or more prior to the Screening Visit. No immunotherapy injections may be received within 48 hours prior to a ragweed pollen exposure visit.
* Non-vaccinated exposure to or active infection with chickenpox or measles within the 21 days preceding the Screening Visit.
* Exposure to systemic corticosteroids for any indication, chronic or intermittent (e.g., arthritis), during the 60 days preceding the Screening Visit, or presence of an underlying condition that can reasonably be expected to require treatment with corticosteroids during the course of the study.
* Use of topical corticosteroids in concentrations in excess of 1% hydrocortisone or equivalent for dermatological conditions within 30 days prior to the Screening Visit
* History of epilepsy or seizures
* History of coronary heart disease, uncontrolled hypertension, or other clinically significant cardiovascular disease.
* Have any of the following conditions that are judged by the investigator to be clinically significant and/or affect the patient's ability to participate in the clinical trial:

  * Impaired hepatic function including alcohol related liver disease or cirrhosis
  * History of ocular disturbances (e.g., glaucoma or posterior subcapsular cataracts)
  * Any systemic infection
  * Hematological, renal, endocrine (except for controlled diabetes mellitis or postmenopausal symptoms or hypothyroidism)
  * Gastrointestinal disease
  * Malignancy (excluding basal cell carcinoma)
  * A current neuropsychiatric condition with or without drug therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Score | 15 mins, 30 mins, 45 mins, 60 mins, 90 mins, 120 mins, and then every hour up to 10 hours post dose

SECONDARY OUTCOMES:
Onset of action of active treatments as compared to placebo | 15 mins, 30 mins, 45 mins, 60 mins, 90 mins, 120 mins and then every hour up to 10 hours post dose
Compare the tolerance as measured by subject questionnaire and adverse events of Captisol-Enabled Budesonide nasal solution, Rhinocort Aqua and Placebo | 15 mins, 30 mins, 45 mins, 60 mins, 90 mins, 120 mins, and then every hour up to 10 hours post dose
Compare the effect and of the three treatments on an EEC-Specific Quality of Life questionnaire | -0.75, 2, 6 and 10 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, MD, Principal Investigator — Allied Research International - Cetero Research
Locations (1):
- Allied Research International - Cetero Research, Mississauga, Ontario, Canada